CLINICAL TRIAL: NCT05380453
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multicenter Trial to Investigate the Efficacy and Safety of Subcutaneously Administered Secukinumab in Patients With New-onset of Giant Cell Arteritis (GCA) Who Are in Clinical Remission and Eligible for Treatment With Glucocorticoid-monotherapy
Brief Title: Efficacy and Safety of Secukinumab in Patients With New Onset of Giant Cell Arteritis Who Are in Clinical Remission
Acronym: GigAINt
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457R1DE01; 2021-002622-24 (EudraCT Number)
Record Dates: First submitted 2022-02-22; First posted 2022-05-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis; GCA; Vasculitis; Vascular Diseases; Secukinumab; Subcutaneous; Vessel Inflammation; Polymyalgia Rheumatica; Arteritis
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis; Vascular Diseases; Polymyalgia Rheumatica; Arteritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo as subcutaneous (s.c.) injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter.
  Interventions: Drug: Placebo to match Secukinumab, s.c.
- Secukinumab (Experimental): Participants will receive secukinumab as subcutaneous (s.c.) injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter.
  Interventions: Biological: Secukinumab 300 mg, s.c.

INTERVENTIONS:
Biological: Secukinumab 300 mg, s.c. — Secukinumab will be administered at a dose of 300 mg as s.c. injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter.
  Other Names: Cosentyx, AIN457
  Arms: Secukinumab
Drug: Placebo to match Secukinumab, s.c. — Placebo will be administered as s.c. injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of subcutaneously (s.c.) administered secukinumab 300 mg in combination with glucocorticoid taper regimen compared to placebo in combination with glucocorticoid taper regimen, in adult patients with new onset of giant cell arteritis (GCA) who are in clinical remission and who are eligible for treatment with glucocorticoid-monotherapy as per current clinical practice and treatment guidelines for the targeted participant population, thereby supporting health technology assessments (HTAs) of secukinumab in Germany.

DETAILED DESCRIPTION:
Recent scientific evidence identified an association between polymorphisms within the IL-17A locus and GCA, supporting a role for IL-17A in vasculitis pathophysiology. Analysis of the inflammatory processes in the aortic wall has indicated that inflammatory cytokines, such as IL-6 and IL-17A are involved in GCA pathogenesis. Elevated IL-17A mRNA levels are correlated with IL-6 and IL-23p19 mRNA levels indicating the involvement of the IL-23/Th17 axis in GCA. With its pleiotropic activity on many different cell types, IL-17A may actively contribute to the inflammatory processes in GCA. In addition, animal studies also support a role of IL-17A as a driver of vasculitis, since mice deficient in IRF-4 binding protein, which have increased IL-21 and IL-17A expression, spontaneously develop arthritis-like joint disease and large vessel vasculitis (LVV).

As secukinumab has already demonstrated a positive benefit/risk profile in the treatment of multiple chronic inflammatory diseases, including PsO, PsA and axSpA, and based on the scientific rationale for targeting the IL-17 pathway in GCA as well as on the basis of the currently ongoing Phase 2 Proof-of-Concept trial the which evaluates the efficacy, safety and tolerability of 300 mg secukinumab compared to placebo, in combination with a 26-week prednisolone taper regimen in adult subjects with GCA (EudraCT number: 2018-002610-12) (Venhoff, et al., 2021), inhibition of IL-17A by secukinumab has a potential therapeutic benefit for GCA patients.

The purpose of this study is to demonstrate the efficacy and safety of subcutaneously (s.c.) administered secukinumab 300 mg in combination with glucocorticoid taper regimen compared to placebo in combination with glucocorticoid taper regimen, in adult patients with new onset of giant cell arteritis (GCA) who are in clinical remission and who are eligible for treatment with glucocorticoid-monotherapy as per current clinical practice and treatment guidelines for the targeted participant population, thereby supporting health technology assessments (HTAs) of secukinumab in Germany.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Participant must be able to understand and communicate with the investigator and comply with the requirements of the study.
3. Male or female participants at least 50 years of age.
4. Diagnosis of new-onset GCA, defined as GCA diagnosed within 6 weeks of baseline (BSL) visit, based on meeting all of the following criteria:

   * Age at onset of disease ≥50 years.
   * History of Erythrocyte Sedimentation Rate (ESR) ≥30 mm/hr or C-reactive protein (CRP) ≥10 mg/L attributable to active GCA.
   * Unequivocal cranial symptoms of GCA (new-onset localized headache, scalp or temporal artery tenderness, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication) AND/OR symptoms of polymyalgia rheumatica (PMR, defined as shoulder and/or hip girdle pain associated with inflammatory morning stiffness) AND/OR symptoms of limb ischemia (claudication).
   * Temporal artery biopsy revealing features of GCA AND/OR evidence of vasculitis in cranial or extracranial arteries by angiography or cross-sectional imaging study such as ultrasound, magnetic resonance angiography (MRA), computed tomography angiography (CTA), positron emission tomography - computed tomography (PET-CT)
5. Participants must be in clinical remission at BSL:

   - Definition of clinical remission: absence of signs and symptoms attributable to active GCA as determined by the investigator.
6. Participants with no relapsing GCA at BSL:

   - Definition of relapsing GCA: occurrence of clinical relapse after clinical remission.
7. Prednisolone or equivalent dose (oral) of 20-60 mg/day or equivalent dose of other glucocorticoids (GCs) at BSL.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study.

3. Participants not eligible for glucocorticoid monotherapy due to known increased risk for or presence of GC-related adverse-effects or complications and/or intolerance to GCs, such as osteoporosis, diabetes mellitus, cardiovascular disease and glaucoma as assessed at the investigator's discretion (see Appendix 15.2).

4. Previous exposure to secukinumab or another biologic drug directly targeting IL-17 or IL-17 receptor.

5. Participants treated with any cell-depleting therapies including but not limited to anti- CD20 or investigational agents (e.g., anti-CD3, anti-CD4, anti-CD5 or anti-CD19).

6. Previous participation in clinical trials for GCA 7. Participants who have been treated with inhibitors directly targeting IL-12 and/or IL-23 (such as ustekinumab, guselkumab, tildrakizumab, risankizumab), IL-1 or IL-1 receptor (such as anakinra or canakinumab), or abatacept within 4 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL.

8. Treatment with tocilizumab, other IL-6/IL6-R inhibitor or JAK inhibitor within 12 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL, or if participant did not respond to or experienced a clinical relapse during treatment any time before BSL.

9. Any treatment received for GCA other than GCs and participant did not respond to treatment or experienced a clinical relapse during treatment any time before BSL.

10. Any other biologics within 4 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL.

11. Participants treated with i.v. immunoglobulins or plasmapheresis within 8 weeks prior to BSL.

12. Participants treated with cyclophosphamide, tacrolimus, everolimus hydroxychloroquine, cyclosporine A, azathioprine, sulfasalazine, mycophenolate mofetil within 6 months prior to BSL.

13. Participants treated with methotrexate (MTX), within 4 weeks prior to BSL. 14. Participants treated with leflunomide within 8 weeks prior to BSL unless a cholestyramine washout has been performed in which case the participant must be treated within 4 weeks of BSL.

15. Participants treated with an alkylating agent within 5 years prior to Baseline, unless specified in other exclusion criteria.

16. Participants requiring systemic chronic glucocorticoid therapy for any other reason than GCA at Screening.

17. Receipt of > 100 mg daily intravenous methylprednisolone pulse therapy within 6 weeks prior to BSL.

18. Participants requiring chronic (i.e., not occasional "prn") high potency opioid analgesics for pain management.

19. Participants treated with any investigational agent within 4 weeks or within 5 half-lives of the drug (whichever is longer) prior to BSL.

20. Contraindication or hypersensitivity to secukinumab. 21. Active ongoing inflammatory diseases other than GCA that might confound the evaluation of the benefit of secukinumab therapy, including inflammatory bowel disease or uveitis.

22. Active ongoing diseases which in the opinion of the investigator immunocompromises the participant and/or places the participant at unacceptable risk for treatment with immunomodulatory therapy.

23. Active ongoing inflammatory diseases or underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions, which in the opinion of the investigator immunocomprises the participant and/or places the participant at unacceptable risk for participation in an immunomodulatory therapy.

24. Major ischemic event (e.g., myocardial infarction, stroke, etc.) or transient ischemic attack (TIA) (except ischemia-related vision loss), related or unrelated to GCA, within 12 weeks of screening.

25. Confirmed diagnosis of any primary form of systemic vasculitis, other than GCA.

26. Active systemic infections during the last 2 weeks (exception: common cold) prior to BSL.

32. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Plus test. Participants with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the participant has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment according to local country guidelines must be initiated prior to BSL.

35. Live vaccinations within 6 weeks prior to BSL or planned live vaccination during study participation until 12 weeks after last study treatment administration.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Time from baseline to first Giant cell arteritis (GCA) clinical relapse | Time from baseline to first GCA clinical relapse, assessed at least up to Week 24
  To demonstrate the superiority of secukinumab 300 mg s.c. compared to placebo (both arms in combination with a prednisolone or equivalent taper regimen as per treatment guideline) in delaying the time to first GCA clinical relapse from baseline in participants with new onset of GCA who are in clinical remission and eligible for treatment with glucocorticoid-monotherapy.
  GCA clinical relapse is defined as both:
  1. The recurrence of signs or symptoms attributable to active GCA after clinical remission, which are considered clinically significant by the investigator AND
  2. The requirement of a change in the treatment prompted by the recurrence of signs and symptoms i. an increase in prednisolone or equivalent dose AND/OR ii. the addition of a rescue treatment.
  Definition of clinical remission: absence of signs and symptoms attributable to active GCA as determined by the investigator.

SECONDARY OUTCOMES:
Proportion of participants in sustained clinical remission at Week 52 | Baseline until Week 52
  To demonstrate the superiority of secukinumab 300 mg s.c. compared to placebo, measured by the proportion of participants in sustained clinical remission at Week 52.
  Definition of sustained clinical remission: absence of signs and symptoms attributable to active GCA between BSL until Week 52.
Changes from Baseline to Week 52 in disease activity and quality of life for the PGA score (VAS) | Baseline to Week 52
  To assess the effect of secukinumab compared to placebo measured by disease activity and quality of life measures at Week 52 for patient global assessment (PGA) of disease activity using a visual analogue scale (VAS)
Changes from Baseline to Week 52 in disease activity and quality of life for the SF-36 (PCS and MCS) score | Baseline to Week 52
  To assess the effect of secukinumab compared to placebo measured by disease activity and quality of life measures at Week 52 for Short form 36 (SF-36 PCS and MCS)
Changes from Baseline to Week 52 in disease activity and quality of life for Patient assessment of pain (NRS) | Baseline to Week 52
  To assess the effect of secukinumab compared to placebo measured by disease activity and quality of life measures at Week 52 for patient assessment of pain using a numeric rating scale (NRS)
Time from Baseline to reach prednisolone or equivalent dose below ≤7.5 mg/day | Baseline to Week 52
  Time to reach prednisolone or equivalent dose below Cushing threshold of ≤7.5 mg/day
Proportion of participants on prednisolone or equivalent dose below Cushing threshold of ≤7.5 mg/day | Bseline to Week 52
  Proportion of participants on prednisolone or equivalent dose below Cushing threshold of ≤7.5 mg/day
Cumulative prednisolone or equivalent dose | Baseline through Week 52
  Cumulative prednisolone or equivalent dose through Week 52
Number of participants with Adverse Events | Baseline up to 52 weeks
  Safety and tolerability assessments over time: incidence and severity of AEs and SAEs; routine safety laboratory parameters
  To evaluate safety and tolerability of secukinumab 300 mg s.c. in participants with new-onset of GCA who are eligible for treatment with glucocorticoid-monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Germany (22):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Bad Abbach
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Sendenhorst
  - Novartis Investigative Site, Trier

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com